CLINICAL TRIAL: NCT07021599
Title: Artificial Intelligence Versus Sonographer Echocardiogram Analysis and Reporting in Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: Artificial Intelligence Versus Sonographer Echocardiogram Analysis and Reporting in Patients With Heart Failure
Acronym: AISEARHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinincal Assistant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2024.587
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Echocardiogram; Artificial Intelligence; Alogrithm; Echocardiological image analysis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored AI echocardiogram analysis and reporting system (Experimental): An experienced cardiologist will be provided with AI's measurements, draft disease grading and report for review. The experienced cardiologist will provide a final grading of left ventricular function, AS and MR on the standardized grading chart, and endorse the final echocardiogram report.
  Interventions: Diagnostic Test: Tailored AI echocardiogram analysis and reporting system
- Echocardiologist interpretation and analysis of Echo images (Active Comparator): An experienced cardiologist (with American Society of Echocardiography level III capacity), will be provided with sonographer's measurements, draft disease grading and report for review.
  Interventions: Diagnostic Test: Tailored AI echocardiogram analysis and reporting system

INTERVENTIONS:
Diagnostic Test: Tailored AI echocardiogram analysis and reporting system — In the AI analysis and reporting pathway, sonographers only need to acquire the echocardiogram images, then the AI algorithm will complete the analysis and report drafting for final endorsement by experienced cardiologists. To ensure blinding of group assignment to the endorsing experienced cardiologists, measurement format and reporting phrases and interface used by AI and sonographers will be standardized.

SUMMARY:
This is a non-inferiority, three-year, multicenter, double-blinded randomized controlled study of an AI versus experienced sonographer echocardiogram analysis in HF patients. Consecutive patients presented for echocardiogram examination with new or worsening HF symptom and positive HF blood markers will be recruited. A target of 514 patients will be randomized 1:1 to receive either AI or sonographer echocardiogram analysis. The primary endpoint of diagnostic accuracy is the complete agreement of disease grading with an experienced cardiologist (American Society of Echocardiography level III) using a standardized grading chart. Important secondary endpoints include the time used for echocardiogram report drafting and report endorsement, 6-month heart failure symptom and hospitalization, and the cost-effectiveness of AI to increase echocardiogram service. Clinical, biochemical and echocardiographic predictors of worsening of heart failure and hospitalization will be identified.

DETAILED DESCRIPTION:
Background Unmet Need for Streamlined Echocardiogram Algorithm Heart failure (HF) is a global pandemic affecting more than 64 million people in the world.

In Hong Kong, the prevalence of HF is estimated to be 2-3% with a steep rise of new onset HF hospitalization in the older age group. The estimated annual worldwide economic burden of HF was 108 billion United States dollars, with direct costs to healthcare systems accounted for 60% and indirect costs to society driven by premature mortality, morbidity and lost productivity accounted for the remaining 40%. Timely diagnosis of HF etiology with early appropriate treatment are critical to reduce HF hospitalization and mortality. While HF with reduced ejection fraction (HFrEF) and preserved ejection fraction (HFpEF) requires different guideline directed medical therapy (GDMT), HF patients with severe valvular heart disease requires interventional treatment. Echocardiogram (cardiac ultrasound) is the key diagnosticmodality to phenotype HF and to guide subsequent appropriate treatment. Access to echocardiogram in Asia Pacific is severely limited (e.g. average waiting time in Hong Kong for routine echocardiogram is 12-18 months), which results in delay in appropriate treatment and hence poor outcomes. While image acquisition is easier to teach, analysis in echocardiogram is time consuming and requires years of training to become proficient, and yet has significant inter-observer variability. Therefore, there is a shortage of fully trained sonographers globally. A streamlined echocardiogram analysis pathway that can enhance the efficiency while improving the diagnostic accuracy of HF etiology is appealing.

Emerging role of Artificial Intelligence in Echocardiogram Artificial intelligence (AI) has emerged as a useful tool with the potential to enhance cardiovascular care including in disease diagnosis, treatment guidance and outcome prediction. Collaborator of this study, David Ouyang et al., has developed machine learning algorithm for fully automated assessment of left ventricular ejection function (LVEF), aortic valve stenosis (AS) and mitral valve regurgitation (MR), with similar accuracy compared to manual analysis by experienced sonographers with reference to cardiologists ("gold standard"). Similar works has also been done by other teams. However, most of these validation studies are conducted based on retrospective echocardiogram cohort. Besides, there can be bias when a different sonographer than the scanning sonographer interprets the images, and that potentially compromised the real-life diagnostic accuracy of sonographers.

Local Heart Failure Data and Application Artificial Intelligence in Echocardiogram Studies from our team has demonstrated that early diagnosis and intensified HF GDMT can reduce HF hospitalization from 13.1% to 8.6% (Hazard ratio = 0.65, p<0.01). Besides, a strong association of 30-day unplanned HF hospitalization with severe valvular heart disease, mostly AS or MR, was found (Odd ratio =72.04, p=0.03). This implies that early phenotyping the mechanism of HF is important. From our unpublished pilot data of patients presented with HF symptom, echocardiogram image acquisition took only 54.2% of the total echocardiogram process time while the remaining were used for analysis by sonographer. When compared, AI used a significantly shorter time for echocardiogram analysis (324 seconds vs 1057 seconds, p<0.01), with a 91.6% agreement rate on LVEF grading and severity of AS and MR. However, this pilot data was collected retrospectively, and the sample size was small. Therefore, it remains unclear whether AI is as accurate and more efficient than experienced sonographers in analyzing multiple possible echocardiogram abnormalities that can interact with each other for HF patients. Moreover, whether the addition of AI analysis will affect the final grading by cardiologists has not been studied.

In this research project proposal, Investigator aim to assess whether a tailored AI echocardiogram analysis and reporting system is as accurate as an experienced sonographer in HF patients by conducting a multicenter double-blinded randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Has new or worsening of heart failure symptoms
* Elevated heart failure blood markers (N-terminal prohormone of brain natriuretic peptide, "NTproBNP") within 3 months from enrolment or by point-of-care blood test, to ensure that the patient's symptoms are cardiac origin
* Provision of written informed consent

Exclusion Criteria:

* Known severe valvular heart disease
* Prior prosthetic valve implantation
* Previously known or suspected >=severe tricuspid regurgitation, >=moderate aortic regurgitation, >=moderate mitral stenosis or pericardial disease during detected during image acquisition
* Insufficient image quality for proper analysis determined by the scanning sonographer (estimated to be 15% of all echocardiograms screened)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-03 (Estimated); Study Completion 2028-12-03 (Estimated)

PRIMARY OUTCOMES:
Rate of complete agreement in LVEF assessments | 6 month
  To assess the rate of agreement in LVEF assessments between AI and sonographers with final adjudication by experienced cardiologist
Rate of complete agreement in assessments of AS severity | 6 month
  To assess the rate of agreement in severity of AS assessments between AI and sonographers with final adjudication by experienced cardiologist
Rate of complete agreement in assessment of MR severity | 6 month
  To assess the rate of agreement in severity of MR assessments between AI and sonographers with final adjudication by experienced cardiologist

SECONDARY OUTCOMES:
Time used for image acquisition echocardiogram process | 6 month
  Compare the time used by AI system and sonographers for image acquisition.
Time used forreport drafting echocardiogram process | 6 month
  Compare the time used by AI system and sonographers for report drafting.
Time used for report endorsement | 6 month
  Compare the time used by AI system and sonographers for report endorsement.
Time used for total echocardiogram process | 6 month
  Compare the time used by AI system and sonographers for total echocardiogram process.
NYHA classification | 6 month
  Compare of NYHA classification of subjects at 6 month and baseline between 2 intervention groups
Symptom burden | 6 month
  Compare of symptom burden of subjects at 6 month and baseline between 2 intervention groups
NTproBNP level | 6 month
  Compare of NTproBNP level of subjects at 6 month and baseline between 2 intervention groups
Rate of heart failure hospitalisation | 6 month
  Compare of Rate of heart failure hospitalisation of subjects at 6 month and baseline between 2 intervention groups
Rate of all-cause mortality | 6 month
  Compare of Rate of all-cause mortality of subjects at 6 month and baseline between 2 intervention groups
Dosage of GDMT | 6 month
  Compare GDMT dosage change of Heart Failure subjects at 6 month and baseline between 2 intervention groups
Rate of valvular intervention | 6 month
  Compare Rate of valvular intervention in subjects with severe valvular heart disease at 6 month and baseline between 2 intervention groups
Rate of LVEF assessment change made by cardiologist on AI generated reports | 6 month
  Rate of LVEF assessment change made by cardiologist on AI generated reports
Rate of change in severity of AS made by cardiologist on AI generated reports | 6 month
  Rate of change in severity of AS made by cardiologist on AI generated reports
Rate of change in severity of MR made by cardiologist on AI generated reports | 6 month
  Rate of change in severity of MR made by cardiologist on AI generated reports
Subgroup analysis of LVEF agreement rate in low complexity disease | 6 month
  To assess the rate of agreement in LVEF assessments between AI and sonographers with final adjudication by experienced cardiologist in low complexity disease
Subgroup analysis of LVEF agreement rate in intermediate complexity disease | 6 month
  To assess the rate of agreement in LVEF assessments between AI and sonographers with final adjudication by experienced cardiologist in intermediate complexity disease
Subgroup analysis of LVEF agreement rate in high complexity disease | 6 month
  To assess the rate of agreement in LVEF assessments between AI and sonographers with final adjudication by experienced cardiologist in high complexity disease
Subgroup analysis of severity of AS agreement rate in low complexity disease | 6 month
  To assess the rate of agreement in severity of AS between AI and sonographers with final adjudication by experienced cardiologist in low complexity disease
Subgroup analysis of severity of AS agreement rate in intermediate complexity disease | 6 month
  To assess the rate of agreement in severity of AS between AI and sonographers with final adjudication by experienced cardiologist in intermediate complexity disease
Subgroup analysis of severity of AS agreement rate in high complexity disease | 6 month
  To assess the rate of agreement in severity of AS between AI and sonographers with final adjudication by experienced cardiologist in high complexity disease
Subgroup analysis of severity of MR agreement rate in low complexity disease | 6 month
  To assess the rate of agreement in severity of MR between AI and sonographers with final adjudication by experienced cardiologist in low complexity disease
Subgroup analysis of severity of MR agreement rate in intermediate complexity disease | 6 month
  To assess the rate of agreement in severity of MR between AI and sonographers with final adjudication by experienced cardiologist in intermediate complexity disease
Subgroup analysis of severity of MR agreement rate in high complexity disease | 6 month
  To assess the rate of agreement in severity of MR between AI and sonographers with final adjudication by experienced cardiologist in high complexity disease

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong